CLINICAL TRIAL: NCT06958432
Title: Node-Sparing Short-Course Radiotherapy Plus Sequential Chemotherapy and PD-1 Inhibitor for Mid/Low pMMR/MSS Rectal Cancer: An Open-Label, Randomized, Prospective Phase II/III Trial (MODIFI-RC-II)
Brief Title: Node-Sparing Short-Course Radiotherapy Sequential Chemotherapy and PD-1 Inhibitor for Mid/Low pMMR/MSS Rectal Cancer (MODIFI-RC-II)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanxin Luo,MD, MD PHD, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025ZSLYEC-417
Record Dates: First submitted 2025-04-24; First posted 2025-05-06 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Rectal Cancer; Neoadjuvant Therapies; Immune Checkpoint Therapy; Radiotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Drug Therapy; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Node-sparing radiotherapy Group (Experimental): Node-sparing short-course radiotherapy followed by sequential chemotherapy and PD-1 inhibitor as total neoadjuvant therapy
  Interventions: Combination Product: Node-Sparing Radiotherapy plus Chemotherapy and PD-1 inhibitor
- Conventional Group (Active Comparator): Conventional short-course radiotherapy followed by sequential chemotherapy as total neoadjuvant therapy
  Interventions: Combination Product: Conventional Radiotherapy plus Chemotherapy and PD-1 inhibitor

INTERVENTIONS:
Combination Product: Node-Sparing Radiotherapy plus Chemotherapy and PD-1 inhibitor — Patients will receive node-sparing modified short-course radiotherapy, followed by six cycles of CAPOX chemotherapy combined with a PD-1 inhibitor. After neoadjuvant treatment, patients will either undergo total mesorectal excision (TME) surgery or enter a watch-and-wait strategy based on clinical assessment.
  Arms: Node-sparing radiotherapy Group
Combination Product: Conventional Radiotherapy plus Chemotherapy and PD-1 inhibitor — Patients will receive conventional-target short-course radiotherapy, followed by six cycles of CAPOX chemotherapy. After neoadjuvant treatment, patients will either undergo TME surgery or enter a watch-and-wait strategy based on clinical assessment.
  Arms: Conventional Group

SUMMARY:
Most rectal cancers are microsatellite stable (MSS) or mismatch repair-proficient (pMMR) and respond poorly to PD-1 inhibitors. Radiotherapy can enhance tumor antigen release and improve responsiveness to PD-1 blockade in MSS/pMMR rectal cancer. Tumor-draining lymph nodes (TDLNs) are critical sites for anti-tumor immune activation, but radiation-induced damage and fibrosis may impair lymphatic drainage and immune responses. Previous studies have reported a remarkable pathologic complete response (pCR) rate of 77.8% using node-sparing radiotherapy in locally advanced rectal cancer. This study aims to evaluate whether node-sparing short-course radiotherapy followed by sequential chemotherapy and PD-1 blockade can improve complete response rate in the phase II part and event-free survival in phase III part, together with sphincter preservation, treatment tolerance, and prognosis in patients with mid-low pMMR/MSS rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* • Voluntarily signs a written informed consent form.

  * Aged between 18 and 75 years at the time of enrollment.
  * Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
  * Expected survival of more than 2 years.
  * Histologically confirmed rectal adenocarcinoma.
  * Tumor biopsy indicates proficient mismatch repair (pMMR), defined by positive immunohistochemical staining for MSH1, MSH2, MSH6, and PMS2, or molecular testing confirms microsatellite stability (MSS).
  * Clinical stage T3-4N0M0 or TanyN+M0 based on the 8th edition of the AJCC TNM classification, as evaluated by high-resolution MRI ± endoscopic ultrasound/transrectal ultrasonography, with the tumor located in the mid-to-lower rectum below the peritoneal reflection.
  * Prior to enrollment, a qualified surgical attending physician must assess the patient's medical history and confirm eligibility for curative R0 resection.
  * No prior systemic or local anti-tumor treatment for rectal cancer, including radiotherapy, chemotherapy, immunotherapy, biologics, or small-molecule targeted therapy.
  * Agrees to provide tumor tissue and peripheral blood samples during screening and throughout the study for research purposes.
  * Adequate organ function, defined as follows:
  * Hematologic (without use of blood components or growth factors within 7 days prior to treatment initiation):
  * Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L
  * Platelet count ≥ 100 × 10⁹/L
  * Hemoglobin ≥ 90 g/L
  * Renal:
  * Calculated creatinine clearance (CrCl) ≥ 50 mL/min using the Cockcroft-Gault formula:

CrCl (mL/min) = [(140 - age) × weight (kg) × 0.85 (if female)] / (72 × serum creatinine [mg/dL])

* Urine protein < 2+ on dipstick or < 1.0 g per 24-hour collection
* Hepatic:
* Total bilirubin ≤ 1.5 × ULN
* AST and ALT ≤ 2.5 × ULN
* Serum albumin ≥ 28 g/L
* Coagulation:
* INR and APTT ≤ 1.5 × ULN
* Cardiac:
* Left ventricular ejection fraction (LVEF) ≥ 50%
* Women of childbearing potential must have a negative urine or serum pregnancy test within 3 days prior to initiating study treatment. If the urine test is inconclusive, a serum test must confirm the negative result. Women of childbearing potential who are sexually active with non-sterilized male partners must agree to use highly effective contraception from screening through 120 days after the last dose of study drug. The need for continued contraception beyond this period should be discussed with the investigator.
* Women of childbearing potential are defined as those who are not surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) and have not undergone menopause (defined as ≥12 months of amenorrhea without alternative medical cause, with FSH levels in the postmenopausal range).
* Highly effective contraception methods are those with <1% failure rate per year when used consistently and correctly (e.g., hormonal contraceptives). In addition to barrier methods, hormonal contraception is required. Periodic abstinence and the calendar method are not considered acceptable.
* Willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study requirements.

Exclusion Criteria:

* • Presence of suspected metastatic lesions or unresectable locally advanced disease, regardless of clinical stage.

  * History of any other malignancy within 5 years prior to enrollment, excluding those considered cured by local therapy (e.g., basal cell carcinoma, squamous cell carcinoma of the skin, superficial bladder cancer, or ductal carcinoma in situ of the breast).
  * Lesions initially staged as T1N0 eligible for local excision, or T2N0 suitable for sphincter-preserving surgery after multidisciplinary discussion.
  * Evidence of acute conditions requiring emergency surgery, such as bowel obstruction, perforation, or gastrointestinal bleeding.
  * Synchronous multiple primary rectal cancers.
  * History of pelvic or abdominal radiotherapy.
  * Inability to swallow tablets, malabsorption syndrome, or any condition affecting gastrointestinal absorption.
  * Prior systemic or local anti-tumor therapy for locally advanced rectal cancer, including curative surgery, chemotherapy, radiotherapy, immunotherapy (e.g., immune checkpoint inhibitors, agonists, or cell-based therapies), biologics, or small-molecule targeted therapy.
  * Use of nonspecific immunomodulatory treatments (e.g., interleukins, interferons, thymic peptides, tumor necrosis factor) within 2 weeks prior to study treatment (excluding IL-11 for thrombocytopenia), or use of herbal or traditional Chinese medicines with anti-tumor indications within 1 week prior to treatment.
  * Active autoimmune disease requiring systemic treatment (e.g., with disease-modifying drugs, corticosteroids, or immunosuppressants) within the past 2 years. Replacement therapies (e.g., thyroid hormone, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency) are not considered systemic treatments.
  * History of or current interstitial lung disease or non-infectious pneumonitis requiring systemic corticosteroid treatment.
  * History of bleeding disorders or coagulopathy; patients requiring long-term anticoagulation (e.g., atrial fibrillation with CHADS2 score ≥ 2).
  * Uncontrolled comorbidities, including but not limited to: decompensated cirrhosis, nephrotic syndrome, uncontrolled metabolic disorders, severe peptic ulcer or gastritis, or psychiatric/social conditions affecting compliance or consent.
  * History of myocarditis, cardiomyopathy, or malignant arrhythmias; unstable angina, heart failure requiring hospitalization, or vascular disease (e.g., aortic aneurysm requiring repair or deep vein thrombosis) within 12 months prior to study treatment; other cardiac conditions impacting safety (e.g., poorly controlled arrhythmia, myocardial infarction, or ischemia).
  * Within 6 months prior to treatment: history of gastroesophageal varices, severe ulcers, non-healed wounds, gastrointestinal perforation, fistulas, bowel obstruction, intra-abdominal abscess, or acute GI bleeding.
  * Arterial thromboembolism, grade ≥3 venous thromboembolism (per NCI-CTCAE v5.0), transient ischemic attack, stroke, hypertensive crisis, or hypertensive encephalopathy within 6 months prior to study treatment.
  * Acute exacerbation of COPD within 1 month prior to treatment; current hypertension not controlled to <160/100 mmHg despite antihypertensive medication.
  * Active or prior inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis) or chronic diarrhea.
  * Severe infections within 4 weeks prior to treatment, including complications requiring hospitalization, sepsis, or severe pneumonia; active infections requiring systemic anti-infective therapy within 10 days prior to treatment (excluding antiviral therapy for HBV or HCV).
  * Major surgery or serious trauma within 30 days prior to treatment; minor local surgery within 3 days (excluding PICC placement).
  * History of immunodeficiency or HIV antibody positivity; long-term systemic corticosteroid or immunosuppressive therapy.
  * Active tuberculosis or suspected TB not ruled out via clinical assessment (e.g., sputum test, chest X-ray); known active syphilis.
  * History of allogeneic organ or hematopoietic stem cell transplantation.
  * Untreated active hepatitis B (HBsAg-positive with HBV DNA > 1,000 copies/mL or 200 IU/mL); active hepatitis C (HCV antibody-positive with detectable HCV RNA).
  * Receipt of a live vaccine within 30 days prior to treatment or planned live vaccination during the study.
  * Known hypersensitivity to any component of the investigational drugs, or history of serious hypersensitivity reactions to monoclonal antibodies.
  * Known history of psychiatric disorders, substance abuse, alcoholism, or drug addiction.
  * Pregnant or breastfeeding women.
  * Any disease, treatment, or abnormal laboratory finding that may interfere with study results, affect full study participation, or is not in the patient's best interest.
  * Systemic or local disease caused by a benign tumor, or tumor-related complications/symptoms that pose high medical risk or survival uncertainty (e.g., leukemoid reaction with WBC > 20 × 10⁹/L, cachexia with >10% weight loss in 3 months prior to screening, or BMI ≤18).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rate | From enrollment to 2 weeks after finishing TNT
  Phase II: Evaluate whether node-sparing modified short-course radiotherapy followed by sequential chemotherapy and PD-1 inhibitor as total neoadjuvant therapy can improve the complete response (CR) rate in mid/low MSS rectal cancer.
Event-Free Survival (EFS) | From enrollment to 3 years after finishing Surgery
  Phase III: To evaluate whether node-sparing modified short-course radiotherapy combined with chemotherapy and a PD-1 inhibitor can improve Event-Free Survival (EFS) in patients with pMMR/MSS rectal cancer.

SECONDARY OUTCOMES:
Sphincter preservation rate | From date of randomization until the date of surgery or the date of watch-and-wait for CR patients，up to 24-30 weeks
Tumor regression grade (TRG) | From enrollment to 2 weeks after finishing TNT
Tumor downstaging rate | From enrollment to 2 weeks after finishing TNT
R0 resection rate | From date of randomization until the date of surgery，up to 24-30 weeks
Incidence of treatment-related adverse events (toxicity) | From enrollment to 2 weeks after finishing TNT
3-year distant metastasis rate | From enrollment to 3 years after finishing Surgery
3-year local recurrence rate | From enrollment to 3 years after finishing Surgery
3-year overall survival (OS) rate | From enrollment to 3 years after finishing Surgery

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No